CLINICAL TRIAL: NCT07064876
Title: A Single-Arm, Phase II Clinical Study of Serplulimab Combined With Cryoablation for Early-Stage Non-Small Cell Lung Cancer
Brief Title: Serplulimab Combined With Cryoablation for Early-Stage Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xi Junjie (Other)
Responsible Party: Sponsor-Investigator, Xi Junjie, Associate Chief Physician, Department of Thoracic Surgery, Zhongshan Hospital Fudan University, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2025098
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Early Lung Cancer
Keywords: Cryoablation; early lung cancer; immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab + Cryoablation (Experimental): Participants in this arm will receive serplulimab combined with CT-guided cryoablation for the treatment of early-stage, inoperable non-small cell lung cancer (NSCLC). Cryoablation will be performed first to locally ablate the tumor. Following recovery, participants will receive intravenous serplulimab at a dose of 300 mg every 3 weeks for up to 6 cycles, starting as soon as no major post-procedural complications are observed. The combination therapy aims to evaluate efficacy (objective response rate) and safety, as well as explore potential biomarkers predictive of treatment outcomes.
  Interventions: Drug: Serplulimab; Procedure: CT-guided Cryoablation

INTERVENTIONS:
Drug: Serplulimab — PD-1 inhibitor, 300 mg intravenous infusion, once every 3 weeks (Q3W) for up to 6 cycles, starting after cryoablation recovery and in the absence of major procedural complications.
Procedure: CT-guided Cryoablation — Percutaneous cryoablation performed under CT guidance to achieve local tumor ablation. Procedure done once (per-protocol) prior to systemic therapy.

SUMMARY:
The goal of this clinical trial is to learn if serplulimab combined with cryoablation can effectively treat early-stage non-small cell lung cancer (NSCLC) in adults who are not eligible for or decline surgery or radiotherapy. The main questions it aims to answer are:

What is the objective response rate (ORR) after combination treatment with serplulimab and cryoablation? What are the progression-free survival (PFS), overall survival (OS), 1-year OS rate, and safety outcomes? This is a single-arm, phase II study with no comparison group.

Participants will:

Receive cryoablation under CT guidance to locally ablate the tumor Receive intravenous serplulimab (300 mg every 3 weeks) for up to 6 cycles Undergo regular imaging and laboratory tests to assess response and monitor safety Provide blood and tissue samples for optional biomarker research The study will enroll 25 patients with stage Ia NSCLC (tumor size >1 cm and ≤3 cm, no ground-glass opacity, EGFR/ALK/ROS1 wild-type) and aims to explore the potential of combining local and systemic immunotherapy in non-surgical candidates.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria to be eligible for the study:

Voluntarily agree to participate in this clinical study. Male or female patients aged ≥18 years at the time of signing the informed consent form (ICF).

Histologically or cytologically confirmed diagnosis of T1N0M0 non-small cell lung cancer (NSCLC) during the cryoablation procedure, classified as stage Ia (tumor size >1 cm and ≤3 cm) according to the 9th edition of the AJCC TNM staging system; patients with ground-glass nodules (GGNs) are excluded.

No detectable driver mutations in EGFR, ALK, or ROS1 genes. Deemed ineligible for or unwilling to undergo surgery or radiotherapy after multidisciplinary team (MDT) discussion.

At least one measurable target lesion within 4 weeks before the first dose, evaluated by the investigator according to mRECIST (2019) criteria.

Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 2. Life expectancy of ≥12 weeks.

Adequate organ function based on laboratory assessments within 14 days before first dose of study treatment, without prior transfusion, albumin, thrombopoietin, or colony-stimulating factor (CSF) support:

Hematologic Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L Platelet count ≥ 75 × 10⁹/L Hemoglobin ≥ 90 g/L Liver function Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) ALT ≤ 5 × ULN AST ≤ 5 × ULN Albumin ≥ 30 g/L Renal function Serum creatinine ≤ 1.5 × ULN; if >1.5 × ULN, creatinine clearance ≥ 50 mL/min (calculated by Cockcroft-Gault formula) Coagulation APTT ≤ 1.5 × ULN PT ≤ 1.5 × ULN INR ≤ 1.5 × ULN Urinalysis Urine protein dipstick ≤ 1+; if ≥ 2+, 24-hour urine protein < 1 g is acceptable Female participants must have a negative serum pregnancy test within 14 days prior to study treatment and agree to use effective contraception during the study and for at least 6 months after the last dose. Breastfeeding is not permitted during the study.

Male participants must agree to use effective contraception or abstain from heterosexual intercourse during the study and for at least 6 months after the last dose. If the male participant has a female partner of childbearing potential or a pregnant partner, he must use condoms to avoid drug exposure to the embryo. Periodic abstinence and withdrawal are not acceptable contraception methods.

Exclusion Criteria:

* Known history of severe hypersensitivity to any monoclonal antibody (Grade >3, per NCI-CTCAE v5.0).

Prior treatment with any immune checkpoint inhibitors, such as anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies.

Known contraindications to cryoablation. Active infection requiring systemic antimicrobial therapy within 14 days prior to the first dose.

History of myocardial infarction within 6 months before first dose, uncontrolled arrhythmias (including QTc ≥450 ms for males or ≥470 ms for females, calculated by Fridericia formula), NYHA Class III or IV heart failure, left ventricular ejection fraction <50%, or clinically significant pleural, pericardial, or peritoneal effusion requiring intervention.

Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, or total serum calcium >12 mg/dL, or corrected calcium >ULN).

History or presence of interstitial lung disease, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or other significant pulmonary conditions that may interfere with evaluation or management of potential treatment-related lung toxicity, as judged by the investigator.

Positive for HBsAg and detectable HBV DNA (active hepatitis B); or positive for HCV antibody and detectable HCV RNA (active hepatitis C); or positive syphilis serology (except non-active infections with specific antibody positive and non-specific antibody negative); or known HIV infection.

Active or suspected autoimmune disease. Patients with stable autoimmune disease not requiring systemic immunosuppressive treatment are allowed.

Active malignancy within 5 years, except for curatively treated localized tumors such as basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, prostate, or breast with ≥5 years disease-free interval.

Receipt of live or attenuated vaccines within 28 days before the first dose or planned during the study. Inactivated seasonal influenza vaccines are allowed.

Receipt of radical radiotherapy within 3 months before the first dose. Presence of spinal cord compression not controlled by surgery and/or radiotherapy.

History of deep vein thrombosis (DVT), ongoing anticoagulant or antiplatelet therapy, or history of severe bleeding or DVT associated with anti-angiogenic therapy.

Poorly controlled hypertension, defined as blood pressure ≥160/100 mmHg despite optimal medical therapy.

Underwent major surgery within 28 days prior to the first dose (major surgery is defined as a procedure requiring at least 3 weeks of recovery before study treatment).

Participation in another interventional clinical trial within 3 months or 5 half-lives (whichever is longer) before screening.

Planned or prior organ or bone marrow transplantation. Known history of psychiatric or substance abuse disorders that may interfere with study compliance or assessments.

Any other condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 12 months
  ORR is defined as the proportion of patients who achieve either a complete response (CR) or partial response (PR) as assessed by investigators using modified Response Evaluation Criteria in Solid Tumors (mRECIST, 2019). Radiological evaluations will be conducted at regular intervals to determine tumor response. The evaluation will be based on measurable target lesions at baseline and follow-up imaging.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 12 months
  PFS is defined as the time from the date of enrollment to the date of disease progression or death from any cause, whichever occurs first. Patients without progression or death will be censored at the last date of tumor assessment.
Overall Survival (OS) | Up to 12 months
  OS is defined as the time from the date of enrollment to the date of death from any cause. Patients alive at the time of analysis will be censored at the date of last follow-up.

OTHER OUTCOMES:
Incidence and Severity of Adverse Events | From first dose to 30 days after last dose of treatment
  Safety will be assessed by the incidence, severity, and relatedness of treatment-emergent adverse events (TEAEs), graded according to CTCAE version 5.0. Laboratory values, vital signs, ECOG performance status, and physical exams will also be monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, No. 180 Fenglin Road, Xuhui District,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided